CLINICAL TRIAL: NCT03689283
Title: The Effect of Dry Needling on Muscle Stiffness, Gait, Motion, and Strength in Healthy Individuals With Latent Trigger Points
Brief Title: The Effect of Dry Needling on Muscle Stiffness, Gait, Motion, and Strength in Healthy Individuals With Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regis University (Other)
Responsible Party: Principal Investigator, Stephanie Albin, Primary Investigator, Regis University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RegisU
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation. Participants in the control group will receive sham needling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental): Individuals in the DN arm will receive two treatment sessions of DN to latent trigger points of the gastrocnemius muscle.
  Interventions: Other: Dry Needling
- Control Group (Sham Comparator): Individuals in the control group will receive two treatment sessions of sham dry needling.
  Interventions: Other: Sham Dry Needlling

INTERVENTIONS:
Other: Dry Needling — Individuals randomized to the Dry Needling Group will receive dry needling to latent trigger points of the gastrocnemius muscle
  Arms: Dry Needling Group
Other: Sham Dry Needlling — Individuals randomized to the Control group will receive sham needling to the gastrocnemius muscle
  Arms: Control Group

SUMMARY:
This study would be the first study to assess the immediate effects of dry needling of latent trigger points of the gastrocnemius muscle on muscle stiffness, gait, range of motion, and strength. The study has the potential to demonstrate that dry needling may have immediate effects on mechanical properties of muscle and may thus guide future treatment for individuals with changes in muscle tissue secondary to pain and/or injury.

DETAILED DESCRIPTION:
Participants will complete the following tests: muscle stiffness testing in both a relaxed and contracted position, GAITRite for spatial and temporal gait characteristics, the Ankle Lunge Test (ALT) to assess range of motion, and calf strength using a dynamometer. Subjects will then receive treatment according to which group they are randomized. Muscle stiffness, gait, motion and strength will be reassessed immediately following treatment at the first session. Four to10 days later, participants will complete the same tests and measures prior to treatment being administered a second time. Another 4-10 days after the second session, participants will complete the tests and measures one final time.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years
2. Able to read and speak sufficient English to complete consent form
3. Symmetrical gait pattern demonstrated through observation
4. Presence of latent trigger point in gastrocnemius muscle

Exclusion Criteria:

1. Any prior foot/ankle surgery, deformity, or injury on the which would affect strength of the gastrocnemius
2. Any prior acupuncture or dry needling within the past month
3. History of systemic disorder in which dry needling would be contraindicated (i.e. bleeding disorders or anticoagulant medication use)
4. Have fractures of the spine, hip, or knee that would likely affect their weight bearing or gait
5. Restrictions in plantar flexion range of motion which would inhibit performing a heel raise
6. No specific calf injury in the past 6 months
7. Participants known or thought to be pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
MyotonPRO | 2 years
  Muscle stiffness will be measured in both a resting and contracted state utilizing this non-invasive device

SECONDARY OUTCOMES:
Knee to wall | 2 years
  Group by time differences will be assessed for talocrural motion (knee to wall)
GAITRite | 2 years
  Group by time differences will be assessed for gait variables (utilizing the GAITRite 6-meter mat)
Handheld dynamometer | 2 years
  Group by time differences will be assessed for strength of the gastrosoleus complex (utilizing a handheld dynamometer)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Albin, PhD, Principal Investigator — Regis University
Locations (1):
- Regis University, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballyns JJ, Turo D, Otto P, Shah JP, Hammond J, Gebreab T, Gerber LH, Sikdar S. Office-based elastographic technique for quantifying mechanical properties of skeletal muscle. J Ultrasound Med. 2012 Aug;31(8):1209-19. doi: 10.7863/jum.2012.31.8.1209. PMID 22837285
- [Background] Bandy WD, Nelson R, Beamer L. COMPARISON OF DRY NEEDLING VS. SHAM ON THE PERFORMANCE OF VERTICAL JUMP. Int J Sports Phys Ther. 2017 Oct;12(5):747-751. PMID 29181252
- [Background] Chuang LL, Wu CY, Lin KC. Reliability, validity, and responsiveness of myotonometric measurement of muscle tone, elasticity, and stiffness in patients with stroke. Arch Phys Med Rehabil. 2012 Mar;93(3):532-40. doi: 10.1016/j.apmr.2011.09.014. Epub 2012 Jan 4. PMID 22222143
- [Background] Furlan AD, van Tulder M, Cherkin D, Tsukayama H, Lao L, Koes B, Berman B. Acupuncture and dry-needling for low back pain: an updated systematic review within the framework of the cochrane collaboration. Spine (Phila Pa 1976). 2005 Apr 15;30(8):944-63. doi: 10.1097/01.brs.0000158941.21571.01. PMID 15834340